CLINICAL TRIAL: NCT05930288
Title: The Role of Short-term Preoperative Walking Exercises in Protecting Cognitive Function and Reducing the Incidence of Surgery-related Complications in the Short Term After Craniotomy in Patients With Supratentorial Brain Tumours
Brief Title: The Effect of Preoperative Walking Exercises on the Prognosis of Supratentorial Brain Tumours Patients After Craniotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202305117
Record Dates: First submitted 2023-06-19; First posted 2023-07-05 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-06

CONDITIONS: Supratentorial Brain Tumor; Exercise; Cognition; Postoperative Complications
MeSH Terms: conditions — Motor Activity; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking exercise (Experimental): Patients receive routine care and exercise as required.
  Interventions: Behavioral: Walking exercise
- Control (No Intervention): Patients receive only routine care.

INTERVENTIONS:
Behavioral: Walking exercise — The target physical activity level for participants is to walk 10,000 steps per day and to meet or exceed that level (but not exceed 15,000 steps) seven days a week for three to four weeks. Participants will be advised to gradually increase their daily step count in proportion to their physical condition. Exercise will be performed by brisk walking or jogging using the indoor treadmill equipped by the Neurosurgery Department of Xiangya Hospital or outdoors. Each workout will begin with a 5-minute warm-up and end with a 5-minute cool-down.
  Arms: Walking exercise

SUMMARY:
The goal of this clinical trial is to learn about in patients with supratentorial brain tumours. The main questions it aims to answer is: Can short-term preoperative walking exercise protect cognitive function in the short term after craniotomy in patients with supratentorial brain tumor and reduce the incidence of surgery-related complications? Participants will be asked to receive general care and regular walking exercises prior to surgery. Researchers will compare patients who receive only general care before surgery to see if preoperative walking exercise has an effect on postoperative prognosis.

ELIGIBILITY:
Inclusion Criteria:

* The participants voluntarily joined this trial and signed the informed consent form, and were able to comply with the research procedures.
* Male and female outpatients or inpatients aged between 18 and 65 years.
* Patients diagnosed with supratentorial tumors through medical history, physical examination, laboratory tests, and head imaging examinations, and without symptoms of intracranial hypertension or epilepsy.
* Patients for elective surgery at low risk, as determined by medical experts based on the patient's actual condition and patient's wishes, who are initially expected to wait for more than three to four weeks before surgery, and for whom, it is anticipated that the condition will not progress during the waiting period.

Exclusion Criteria:

* The patient with a substantial brain tumor who is significantly susceptible to tumor stroke or brain herniation.
* Patients with a clinical diagnosis of cerebral haemorrhage or intracranial infection or epilepsy.
* Patients with acute or unstable heart disease (e.g. unstable angina or severe aortic stenosis).
* Patients with a physical status of Grade 3, 4 or 5 according to the American Society of Anesthesiologists classification.
* Patients with disabling orthopaedic or neuromuscular conditions.
* Patients with a history of clinically diagnosed cognitive impairment, such as dementia and mental retardation.
* Patients with a current or previous diagnosis of significant mental illness, chronic neurological disease or active substance abuse (as per the Diagnostic and Statistical Manual of Mental Disorders 5th edition).
* Patients with heart failure (New York Heart Association Class 3 or Class 4 functional class).
* Patients with severe chronic obstructive pulmonary disease (exertional expiratory volume in the first second of exhalation < 50% of predicted value).
* Patients with anaemia (symptomatic or haematocrit < 30%).
* Patients who have participated in other trials 1 month before or during the trial.
* Patients who are prohibited from exercising without face-to-face supervision as assessed by the Physical Activity Readiness Questionnaire (PAR-Q) or as judged by the exercise physician based on the cardiopulmonary exercise testing (CPET).
* Patients who are unable to cooperate during the Montreal Cognitive Assessment (MoCA) test due to impaired consciousness or mental impairment.
* Patients with motor dysfunctions, such as hemiplegia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative cardiopulmonary complications (pneumonia, thrombosis, etc. [by Japan Clinical Oncology Group postoperative complications criteria]) | 1 week post-operative/discharge (select whichever occurs first)
  Type and number of surgery-related cardiopulmonary complications that occurred after the patient's surgery.
Cognitive function change (by Montreal Cognitive Assessment [MoCA], MoCA Chinese 7.1 and MoCA Chinese 7.2 [both ranging from 0 to 30 points, with higher scores generally indicating better cognitive function]) | Baseline, 14 days preoperatively, three days preoperatively, 1 week post-operative/discharge (select whichever occurs first)
  The gap between patients' post-operative and pre-operative cognitive function. MoCA Chinese 7.1 for baseline and 14 days preoperatively, MoCA Chinese 7.2 for three days preoperatively and 1 week post-operative/discharge (select whichever occurs first).

SECONDARY OUTCOMES:
Average length of stay | Discharge (up to 12 weeks)
  Average length of hospital stay for patients.
Postoperative pain (by 0-10 Numerical Rating Scale [0 to 10 points, with higher scores generally indicating more severe pain]) | 1 week post-operative/discharge (select whichever occurs first)
  Degree of pain felt by patient in the postoperative period.
Subject satisfaction (by Patient Satisfaction Questionnaire-III [50 to 250 points, with higher scores generally indicating higher satisfaction]) | 1 week post-operative/discharge (select whichever occurs first)
  Patient satisfaction with health care provided by physicians.
Cost of care | 1 week post-operative/discharge (select whichever occurs first)
  The researcher will estimate the costs of hospitalisation and interventions based on data from hospital records, with unit costs taken from standard estimated costs from the Office of Medical Pricing. The analysis of program implementation costs will take into account clinician salaries, overheads and equipment costs. Formal care costs will be extracted from medical records and institutional databases, considering preoperative characteristics, type of surgery and postoperative recovery, and any complications.
Incidence of other postoperative surgery-related complications (cerebral haemorrhage, intracranial infections, etc.) | 1 week post-operative/discharge (select whichever occurs first)
  Type and number of other surgery-related complications (cerebral haemorrhage, intracranial infections, etc.) that occurred after the patient's surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fangkun Liu, MD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Due to protect the patients' privacy, the investigators will not make individual patient data (IPD) publicly available. Other researchers intending to obtain IPD may contact the investigators to make a request. The investigators may share IPD if the request is approved by the Ethics Committee.

REFERENCES:
- [Derived] Qu C, Cao Z, Zhou J, He S, Liu F, Liu Z. Preoperative walking exercise to improve prognosis in patients with supratentorial brain tumours after craniotomy: protocol for a randomised controlled trial. BMJ Open. 2024 May 15;14(5):e080787. doi: 10.1136/bmjopen-2023-080787. PMID 38754891